CLINICAL TRIAL: NCT05462886
Title: Clinical Performance of Masimo INVSENSOR00057 for Heart Rate Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1020
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Masimo INVSENSOR00057 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo INVSENSOR00057 device.
  Interventions: Device: Masimo INVSENSOR00057

INTERVENTIONS:
Device: Masimo INVSENSOR00057 — Noninvasive wearable health monitoring device

SUMMARY:
This study is designed to compare the accuracy of a noninvasive measurement of heart rate compared to reference values obtained by a standard of care ECG monitor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 80 years of age.
* Subject is able to read and communicate in English.

Exclusion Criteria:

* Subject has open wounds, inflamed tattoos or piercings on the area of device placement, and/or has any visible healing wounds that the investigator and/or medical professional determines may place them at an increased risk for participation.
* Subject has any medical condition which in the judgment of the investigator and/or study staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Masimo INVSENSOR00057
Started | 86
Completed | 79
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Masimo INVSENSOR00057
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 21
  More than one race | 8
  Unknown or Not Reported | 24
Region of Enrollment [Number; unit: participants]
  United States | 79

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Accuracy of Masimo INVSENSOR00057
Description: Heart rate accuracy was determined by calculating the accuracy root mean-squared (Arms) difference between the measured values from Masimo INVSENSOR00057 (TestHR_i) to the reference ECG monitor values (RefHR_i).
  Arms= √(∑(i=1 to n) ((TestHR_i-RefHR_i )^2 ))/n
Time Frame: 1-3 hours
Population: 17 subjects not included in analysis due to data collection error.
Measure: Number; unit: bpm
Groups:
- INVSENSOR00057: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00057 device.
  INVSENSOR00057: noninvasive wearable health monitoring device
Arm/Group | INVSENSOR00057
Number analyzed (Participants) | 62
bpm | 1.38

ADVERSE EVENTS:
Time Frame: 1-3 hours
Arm/Group | Masimo INVSENSOR00057
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT05462886/Prot_SAP_000.pdf